CLINICAL TRIAL: NCT06097793
Title: KSD-101 Therapy for EBV-associated Nasopharyngeal Carcinoma: an Exploratory Clinical Trial
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Kousai Bio Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSD-101-CR003
Record Dates: First submitted 2023-10-16; First posted 2023-10-24 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: EBV; Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KSD-101 (Experimental): Biological: Dendritic Cell Vaccine（Autologous monocyte-derived DCs pulsed with EBV Multi-antigen).
  Interventions: Biological: KSD-101

INTERVENTIONS:
Biological: KSD-101 — Patients will receive approximately 5x10^6 DC vaccine via subcutaneous injections bi-weekly,total 3-5 times.

SUMMARY:
The main purpse of this study is to evaluate the safety of KSD-101 in patients with EBV-associated Nasopharyngeal Carcinoma,to evaluate the initial clinical outcomes and evaluate the immune response to KSD-101 for the treatment in Patients with EBV-associated Nasopharyngeal Carcinoma

DETAILED DESCRIPTION:
This is a single-center, single-arm, open, multiple-dose clinical study，evaluating the safety, preliminary efficacy, and immune response of KSD-101 for the treatment of patients with EBV-associated nasopharyngeal carcinoma.

Enrolled subjects will receive a peripheral blood single nucleated cell collection (D-20) of approximately 120-150 ml. After the single collection is transported to the dendritic cell vaccine preparation party via the cold chain, a dendritic cell vaccine (KSD-101) will be prepared using the subject's own single nucleated cells. After successful preparation of KSD-101, the subject will return to the hospital for KSD-101 reinfusion as follows.

1. KSD-101 route of administration: subcutaneous injection.
2. KSD-101 treatment dose: 5.0 × 10^6 cells/dose.
3. KSD-101 treatment frequency: once every 2 weeks for a total of 3-5 times. The 4th and 5th times are booster treatments, which need to be decided by the investigator according to the condition of the subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients or their legal guardians voluntarily participate and sign the informed consent form.
2. male or female patients aged 18-70 years (inclusive of the cut-off value) on the date of signing the informed consent.
3. Nasopharyngeal carcinoma confirmed by pathological tissue examination and EBER-positive in tumor tissue by in situ hybridization (ISH or FISH).
4. nasopharyngeal carcinoma with localized recurrence or localized recurrence with systemic metastasis, or primary metastatic nasopharyngeal carcinoma unsuitable for localized or radical treatment, for which there is no effective treatment and which is seriously life-threatening.
5. at least one measurable lesion according to RECIST v1.1 criteria.
6. have an Eastern Cooperative Oncology Group (ECOG) score: 0-1.
7. have criteria for single or venous blood collection and have no other contraindications to cell collection.
8. the patient's laboratory findings are compatible:

   * Blood routine: neutrophils ≥ 1.0×10^9/L, hemoglobin ≥ 80g/L, platelets ≥ 50×10^9/L.
   * Liver function: ALT, AST ≤ 3 × ULN and total bilirubin ≤ 1.5 × ULN.
   * Renal function: creatinine ≤ 1.5 × ULN.
   * Cardiac function: left ventricular ejection fraction (LVEF) ≥ 40%.
   * Coagulation function: fibrinogen ≥ 1.0g/L, activated partial thromboplastin time (APTT) ≤ 1.5 × ULN, prothrombin time (PT) ≤ 1.5 × ULN.
9. The patient's corresponding lymph node region can meet the demand for subcutaneous injection.

Exclusion Criteria:

1. Patients receiving any anti-tumor therapy such as chemotherapy, radiotherapy, immunosuppressive therapy, etc. within 4 weeks prior to mono-collection.
2. Women who are pregnant (positive urine/blood pregnancy test), breastfeeding, or men or women who are planning to conceive within the last 1 year.
3. active hepatitis B (HbsAg or HbcAb positive and HBV DNA ≥100 IU/mL), active hepatitis C (HCV antibody positive and peripheral blood HCV RNA positive); human immunodeficiency virus (HIV) antibody positive; syphilis test positive.
4. patients with central nervous system pathology (e.g., cerebral edema, need for hormonal intervention, or progression of brain metastases).
5. patients with uncontrollable infectious disease within 4 weeks prior to enrollment, or with active tuberculosis or on anti-tuberculosis therapy. (< CTCAE grade 2 genitourinary infections and upper respiratory tract infections, except EBV infections).
6. the patient has a serious underlying disease (cardiovascular disease, respiratory disease, renal insufficiency, coagulation abnormality, autoimmune disease or immunodeficiency disease, etc.).
7. other active malignant tumors within the past 3 years, unless they are curable tumors and have been significantly cured, such as basal or squamous cell carcinoma, carcinoma in situ of the uterine cervix or breast.
8. subjects who have undergone major surgery or severe trauma within 4 weeks prior to enrollment or are expected to require major surgical intervention (i.e., surgery requiring the assistance of endotracheal anesthesia) during the study period.
9. the patient has received a prophylactic live or live attenuated vaccine within 4 weeks prior to screening.
10. the patient has participated in another clinical study within 4 weeks prior to screening.
11. patients with a prior history of severe drug allergy, or penicillin allergy.
12. the patient has substance abuse/addiction.
13. patients with other conditions that, in the judgment of the investigator, make them unsuitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety endpoint | 1 year after DC Vaccines injection
  Adverse events will be graded according to the NCI-CTCAE 5.0 grading criteria throughout the study period, except for injection site (localized) adverse events, which will be graded with reference to the Guidelines for Grading Criteria for Adverse Events in Clinical Trials of Vaccines for Prophylaxis. Monitor and assess the incidence and relevance to study drug and severity of all adverse events, vital signs, physical examination and laboratory findings.

SECONDARY OUTCOMES:
EBV-DNA load | 1 year after DC Vaccines injection
  Antiviral effect: changes in EBV-DNA load were assessed during the study
Objective response rate (ORR) | 1 year after DC Vaccines injection
  The percentage of participants who achieved PR or better response
Disease control rate (DCR) | 1 year after DC Vaccines injection
  The percentage of participants who achieved SD or better response
Duration of response (DOR) | 1 year after DC Vaccines injection
  DOR will be calculated among responders (with a PR or better response) from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease
Progression-free survival (PFS) | 1 year after DC Vaccines injection
  The time from the start of CAR-GPRC5D treatment for the participants to the first time of disease progression or death for any reason
Overall survival (OS) | 1 year after DC Vaccines injection
  OS is measured from the date of the initial injection of DC Vaccines to the date of the participant's death
Levels of EBV-specific CD8+ T cells | 1 year after DC Vaccines injection
  EBV-specific CD8+ T cells in peripheral blood will be assessed to monitor changes
Levels of B cells | 1 year after DC Vaccines injection
  B cells in peripheral blood will be assessed to monitor changes
Levels of NK cells | 1 year after DC Vaccines injection
  NK cells in peripheral blood will be assessed to monitor changes
According to EORTC QLQ-C30 | Up to 1 year
  Changes of Quality of life, according to EORTC QLQ-C30
According to EQ-5D-5L | Up to 1 year
  Changes of Quality of life, according to EQ-5D-5L
According to EORTC QLQ-H&N35 | Up to 1 year
  Changes of Quality of life, according to EORTC QLQ-H&N35
According to ECOG fitness status | Up to 1 year
  Changes of Quality of life, according to ECOG fitness status

CONTACTS AND LOCATIONS:
Overall Officials: Guangyuan Hu, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China